CLINICAL TRIAL: NCT01179906
Title: Effect of Lifestyle Interventions on the Progression of Kidney Disease in Patients With Chronic Kidney Disease
Brief Title: Lifestyle Modifications and the Progression of Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Springfield College (Other)
Collaborators: Western New England Renal & Transplant Associates (Unknown)
Responsible Party: Samuel Headley, Springfield College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BHS research incubator study
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2006-01

CONDITIONS: Patients With Stage 2-4 Chronic Kidney Disease
Keywords: CKD
MeSH Terms: interventions — Exercise; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle intervention-exercise & diet (Experimental): Subjects trained for 48 weeks with a personal trainer
  Interventions: Behavioral: Exercise training; Behavioral: Diet modification

INTERVENTIONS:
Behavioral: Exercise training — Subjects exercise trained for 48 weeks with personal trainers at a college wellness center
Behavioral: Diet modification — Exercise training using personal trainers 3 times per week. Individuals were trained at a moderate intensity

SUMMARY:
Aerobic training has been shown to favorably alter several of the known risk factors for coronary artery disease including hypertension, dyslipidemia, obesity, and diabetes (1). It seems logical that if these risk factors were aggressively controlled in patients with chronic kidney disease (CKD) by implementing lifestyle changes (e.g., diet and exercise training) to support the pharmacologic interventions that are necessary for the control of the disease, then the rate of progression of the disease may be altered. However, to date, there is no clear research evidence to support this hypothesis. Therefore the aims of the proposed study are:

1. To test the hypothesis that lifestyle interventions (i.e., dietary modification and regular, long-term aerobic exercise training) will favorably alter the natural progression of CKD in a sample of patients compared to a control group who will receive the current standard care.
2. To explore possible mechanisms that could contribute to the observed changes.

ELIGIBILITY:
Inclusion Criteria:

* Stages 2-4 CKD

Exclusion Criteria:

* CAD
* MI

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) | 48 weeks
  GFR was estimated using the MDRD equation, creatinine clearance, urea clearance

SECONDARY OUTCOMES:
24 hour urine protein output | 48 weeks
  urine protein output is measured before and after 48 weeks of the training program

CONTACTS AND LOCATIONS:
Overall Officials: Sam A Headley, Ph.D, Principal Investigator — Springfield College
Locations (1):
- Springfield College, Springfield, Massachusetts, United States